CLINICAL TRIAL: NCT06586541
Title: Family Participation in Intensive Care Unit Rounds (The Family-ICU Trial)
Brief Title: The Family-ICU Trial
Acronym: Family-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Michael Goldfarb, Attending Staff, Division of Cardiology, Lady Davis Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2025-4182
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Virtual Care; Family Engagement; Patient and Family Engagement; Health Care Delivery; Family-centered Care; Physician Rounds; Critical Care, Intensive Care
Keywords: Patient- and Family-Centered; Patient- and Family-Centered Care; Family Engagement; Critical Care; Intensive Care Unit; Person-Centered Care; Delivery of Health Care; Virtual Rounds; Family Participation in Rounds; Physician Rounds

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (Control group) (No Intervention): Participants will be able to engage in care as per current family engagement practices. Family members in the usual care group will not participate in daily ICU rounds. In-person or virtual family participation in rounds is not routinely performed at any of the trial sites.
- Phase 2 (Intervention) (Experimental): Participants in the Intervention group will be invited to participate in attending team rounds.
  Interventions: Other: Participation in attending team rounds

INTERVENTIONS:
Other: Participation in attending team rounds — Family members can participate both in-person and virtually, which can vary daily if desired. If the family member wishes to participate in-person, they will be invited to be present when the team rounds in the ICU. If the family member wishes to participate virtually, they will be provided with a personalized link by email to attend rounds.
  Arms: Phase 2 (Intervention)

SUMMARY:
Family inclusion in adult intensive care unit (ICU) rounds is recommended by critical care professional societies, yet widespread uptake of this practice is limited. A key barrier cited by ICU clinicians is insufficient evidence to support this practice. There is a need for robust evidence to support family participation in adult ICU rounds and influence change to routine clinical care. The primary purpose of this study is to assess whether family participation in adult ICU rounds improves family engagement in care. The secondary objectives are to assess family satisfaction, and anxiety and depression, to explore user experiences of family participation in ICU rounds, and to evaluate strategies to improve family member recruitment and retention rates. This is a stepped-wedge cluster randomized trial (n=194) at 6 Canadian ICUs. The stepped wedge cluster randomized trial is a pragmatic study design that overcomes methodological limitations in evaluating a healthcare service delivery intervention. In the stepped-wedge cluster design, there is random and sequential crossover of clusters from control (phase 1) to intervention (phase 2) until all clusters are exposed. The stepped-wedge design also allows each site to function as its own control. The stepped-wedge design is more powerful than a parallel design when substantial cluster level effects are present.

ELIGIBILITY:
Inclusion Criteria:

* Adult family members (age ≥ 18 years) of ICU patients
* Expected ICU stay ≥ 48 hours
* Family members wishing to participate in rounds virtually must have the technological capability and understanding to participate virtually (must have a phone or computer with internet and audio/video capabilities)

Exclusion Criteria:

* Family members who do not wish to participate in care
* Repeat admissions within the study period
* Another family member has already participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
FAMily Engagement (FAME) score within 1 week of ICU discharge | 1-week post-hospital discharge
  The FAMily Engagement (FAME) tool is a self-administered 12-item questionnaire that assesses an individual's current engagement practice. FAME uses a five-point Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree), and scale results are changed to a 0-100 scoring system, with higher scores indicating greater engagement in care. The following subdomains are evaluated: engagement perception, family presence, communication, education, decision-making, care contribution, and family needs. FAME includes the following engagement domains: family presence, family needs, communication and education, decision making, and direct care. FAME also captures the following family-centered care principles: dignity and respect, information sharing, participation, and collaboration.

SECONDARY OUTCOMES:
Quality of communication (QOC score) | 1-week post-hospital discharge
  The Quality of Communication tool is a 13-item questionnaire that was developed and validated in an ICU setting to measure the perceived quality of communication. Scores range from 0 to 100, with higher scores indicating better clinician-family communication.
Anxiety and depression (HADS) | 6 months post-hospital discharge
  The Hospital Anxiety and Depression Scale (HADS) is a simple to use, validated, and widely used self-reported tool to measure anxiety and depression in medical patients. The survey is composed of 14 questions: 7 depression-related and 7 anxiety-related questions. The score for each item ranges from 0 to 3, and subscale scores greater than 8 denotes anxiety or depression.
Anxiety and depression (HADS) | 1-week post-hospital discharge
  The Hospital Anxiety and Depression Scale (HADS) is a simple to use, validated, and widely used self-reported tool to measure anxiety and depression in medical patients. The survey is composed of 14 questions: 7 depression-related and 7 anxiety-related questions. The score for each item ranges from 0 to 3, and subscale scores greater than 8 denotes anxiety or depression.
Post-traumatic stress (IES-Revised) | 6 months post-hospital discharge
  The IES-Revised is a 22-item questionnaire that has been validated and is widely used for measuring post-traumatic stress symptoms and yields a total score ranging from 0 to 88 and subscale scores for the Intrusion, Avoidance, and Hyperarousal subscales. Items are rated on a 5-point scale ranging from 0 (not at all) to 4 (extremely). High scores indicate greater severity of PTSD.
Family satisfaction in the ICU (FS-ICU) | 1-week post-hospital discharge
  The Family Satisfaction in the ICU survey (FS-ICU) is a 24-item instrument that was developed and validated to assess family satisfaction and experience with care in the ICU. Scores range from 0 to 100, with higher scores indicate greater satisfaction.
Quality of life (EuroQOL-5D-5L score) | 6 months post-hospital discharge
  The EuroQOL-5D-5L is a 5-item questionnaire that has been validated and is widely used for measuring health-related quality of life. Each dimension has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The scores are combined to generate a single index value for overall health status. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Goldfarb, MD, MSc, Principal Investigator — Lady Davis Institute, McGill University, Jewish General Hospital
Locations (2):
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No